CLINICAL TRIAL: NCT01014260
Title: Doxycycline Outcomes in Lupus Erythematosus: (DOLE)
Brief Title: Doxycycline Outcomes in Lupus Erythematosus
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: We could not get funding for study.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Michelle Petri, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NA_00001755
Record Dates: First submitted 2009-11-12; First posted 2009-11-16 (Estimated); Last update posted 2012-03-30 (Estimated); Status verified 2010-05

CONDITIONS: Cardiovascular Disease
Keywords: Inflammatory markers of cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Doxycycline

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo
- Doxycycline (Active Comparator): Doxycycline
  Interventions: Drug: Doxycycline

INTERVENTIONS:
Drug: Placebo — This is a randomized double-blind clinical trial of doxycycline 20 mg bid versus 100mg bid versus placebo, given for 3 months, to be conducted at a single center (JHH).
  Arms: Placebo
Drug: Doxycycline — Doxycycline 20 mg bid versus Doxycycline 100 mg bid versus placebo
  Arms: Doxycycline

SUMMARY:
Cardiovascular disease, specifically from atherosclerosis, is the major cause of mortality in SLE in developed countries. In a recent study the investigators have shown that high sensitivity C reactive protein (hs-CRP) is higher in SLE patients with (versus without) coronary calcium, a measure of subclinical atherosclerosis. In an ongoing two year intervention trial of atorvastatin, the investigators will determine if statins retard coronary calcium and reduce hs-CRP. However, 10% of the patients in the trial were intolerant of statins. The investigators want to now investigate whether there are additional, and potentially safer ways, to reduce hs-CRP in SLE. In this study, the investigators will determine if doxycycline reduces hs-CRP and other vascular inflammatory markers including interleukin 6 (IL-6), soluble vascular cell adhesion molecule (sVCAM-1), soluble inter cell adhesion molecule (s-ICAM-1) and matrix metalloproteinase 9 (MMP-9) in SLE.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a clinical diagnosis of SLE, with a hs-CRP above > 3mg/L, (high risk level) for the last 3 months, are eligible.
2. Patients must be 18 years of age or older and able to give informed consent.
3. Contraception other than OCPs is necessary if a woman is at risk for pregnancy.

Exclusion Criteria:

1. SLE patients who are allergic to doxycycline or other tetracyclines.
2. Patients who are pregnant or are planning to become pregnant.
3. Patients who are on oral contraceptives (any method of contraception other than OCPs can be used.
4. Tetracycline use within the previous 2 weeks of enrollment.
5. Patients who are currently on statins will be excluded, because statins might reduce hs- CRP.
6. Patients who are on warfarin.
7. Patients whose most recent EKG shows significant cardiac dysrhythmias or heart block.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-09; Primary Completion 2011-03 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Determine whether doxycycline 20 mg bid (periostat) versus 100mg bid versus placebo is more effective in reducing hs-CRP. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Petri, M.D, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University SOM. 1830 East Monument St, Ste 7500, Baltimore, Maryland, United States